CLINICAL TRIAL: NCT03416205
Title: A Prospective Study of Treating Duodenal Papillary Sphincter in Different Ways During ERCP: Comparison of EST, EPBD, and sEST+EPBD in Endoscopic Choledocholithiasis Treatment.
Brief Title: A Prospective Study of Treating Duodenal Papillary Sphincter in Different Ways During ERCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Zhujiang Hospital (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-XHNK-001
Record Dates: First submitted 2017-05-15; First posted 2018-01-31 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2017-05

CONDITIONS: ERCP

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EST (Experimental): EST is an operation using the Erbao electric knife and Three-cavity incision knife to make a large incision to the duodenal nipples，and the incision scope is the nipple mouth uplift length of 4/5. It has been used since 1974. The technique is intuitive and intact. However, EST cut too small to achieve the purpose of treatment and will affect the next step, and if the incision is too large it may be easier to occur gastrointestinal perforation and bleeding.The EST will also damage the anatomy of the Oddi sphincter structure,which causes bacterial reflux to the bile duct, the recurrence of CBD.Some surgeons prefer it because it's postoperative pancreatitis rate is lower and it may be easier to find the lesion position if bleeding or perforation occurs.
  Interventions: Device: Erbao electric knife; Device: Three-cavity incision knife
- EPBD (Experimental): EPBD is an operation using the Columnar expansion balloon to expand duodenal to achieve the purpose of using the basket and other instruments to take stone out. Balloon expansion may retain part of the sphincter not destroyed, and basically retain the normal physiological function of the nipple sphincter.Thus it may reduce the risk of recurrence of stones and bacterial reflux. However,the postoperative pancreatitis rate is high(4.8% -19.5% ), and nipple sphincter tear is uncontrollable in EPBD.If the digestive tract perforation or bleeding occur after EPBD,it is hard to accurately find the lesion position.Some surgeons prefer it for it's lower bleeding and perforation rate.
  Interventions: Device: Columnar expansion balloon
- sEST+EPBD (Experimental): sEST+EPBD is an operation combining EST and EPBD. Investigators use the Erbao electric knife and Three-cavity incision knife to make a small incision to the duodenal nipples, and the incision length is less than 5mm while the incision scope is less than the nipple mouth uplift length of 1/2. Then, Investigators match the appropriate Columnar expansion balloon according to the diameter of the common bile duct and gradually expand the duodenal nipples.This method allows the nipple sphincter to be cut in a small range, then the balloon can guide the direction of the nipple sphincter tearing after the expansion , so that the digestive tract bleeding, perforation may be smaller and more controllable. Besides,it may reduce postoperative pancreatitis rate and the recurrence rate of stones.
  Interventions: Device: Erbao electric knife; Device: Three-cavity incision knife; Device: Columnar expansion balloon

INTERVENTIONS:
Device: Erbao electric knife — Erbao electric knife is used to cut the Duodenal sphincter
  Arms: EST; sEST+EPBD
Device: Three-cavity incision knife — Three-cavity incision knife is used to cut the Duodenal sphincter
  Arms: EST; sEST+EPBD
Device: Columnar expansion balloon — Columnar expansion balloon is used to expand the the Duodenal sphincter
  Arms: EPBD; sEST+EPBD

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is commonly performed to remove bile duct stones.Endoscopic sphincterotomy (EST), endoscopic papillary balloon dilation (EPBD), and endoscopic sphincterotomy plus balloon dilation (sEST+EPBD) are 3 methods used to enlarge the papillary orifice, but their efficacy and safety remains controversial. This study aimed to compare these methods for treating common bile duct (CBD) stones.

DETAILED DESCRIPTION:
Investigators first divided the patients with different sizes of common bile duct stones into two groups. The bile duct stone diameter of group A is less than 1.0cm while group B is more than 1.0cm and less than 1.5cm. Each group compared Endoscopic sphincterotomy (EST), endoscopic papillary balloon dilation (EPBD), and endoscopic sphincterotomy plus balloon dilation (sEST+EPBD) in ERCP. Through the postoperative comparison of relevant inspection test indicators, the recovery of patients, whether the occurrence of complications, including infection,bleeding,pancreatitis,perforation , and 1 year stone recurrence rate,Investigators assess the advantages and disadvantages in three different strategies in different sizes of common bile duct stones , and finally get a relatively objective evaluation to guide our daily ERCP work on the choice of duodenal papillary sphincter treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-80 years old
* CT or MRCP diagnose the patients with Common bile duct stones
* The diameter of the stone is less than or equal to 1.5cm
* Patients with the indications for ERCP
* Patients and their families agree to participate in the trial

Exclusion Criteria:

* Stones are too large (> 1.5cm)
* A history of gastrointestinal surgery
* ERCP and EST or EPBD surgery history
* Patients generally poor, total bilirubin> 200umol / L or PT time extension> 3s
* Patients with mental illness or other serious heart and lung disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
the incidence of composite events of infection, hemorrhage, perforation, pancreatitis | 3 and 24 hours after the ERCP
  Investigators comprehensively assess whether the hemorrhage, perforation, pancreatitis and other complications of retrograde cholangiopancreatography (ERCP) happen or not by clinical sympton and blood index 1 day after the ERCP. The blood index includes CRP, amylase,lipase,leukocyte,red blood cell,hemoglobin.Besides,CT will be done if necessary.Finally investigators use statistical method to analyse the incidence of composite events of infection, hemorrhage, perforation, pancreatitis.

SECONDARY OUTCOMES:
Recurrence rate of bile duct stones | 1 year after the ERCP.
  One year after the ERCP,the participants will have a CT scan to find out whether the bile duct stones recur again.

CONTACTS AND LOCATIONS:
Overall Officials: Changhui Yu, Doctor, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided